CLINICAL TRIAL: NCT05677945
Title: A Randomized Controlled Trial Comparing the Clinical and Radiographic Success of 3Mixtatin Versus Modified 3Mix in Lesion Sterilization and Tissue Repair (LSTR) for The Treatment of Necrotic Primary Molars
Brief Title: 3Mixtatin Versus Modified 3Mix-MP in Lesion Sterilization and Tissue Repair for Treatment of Necrotic Primary Molars
Acronym: LSTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Magdy Abdel Azeem Al Shamy, Masters Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LSTR in necrotic primary teeth
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Necrotic Primary Molars
Keywords: 3MIX-MP; 3Mixtatin; LSTR
MeSH Terms: interventions — Propylene Glycol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This research will be a double-blinded study, where the patient (participant) and the outcome assessor will be blinded to the treatment group (to avoid detection, reporting and assessment bias).
  When a patient agrees to participate in the trial, an envelope will be drawn by one of the residents present at the clinic and name, telephone number and patient's I.D. will be written on it. Those selected envelops will be opened at treatment visit after performing access cavity to choose which material should be used. Randomization and allocation concealment will be performed by the co-supervisor to avoid selection bias. The participant will not be aware of which treatment modality he will be receiving.
  Principal investigator will not be blinded due to differences in preparation of the mix.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group I Experimental Group):Simvastatin mixed with modified triple antibiotic (3Mixtatin) (Experimental): Patients will then be allocated into either one of the groups alternatively after access cavity preparation depending on the mix to be used as follows:
  for this group:
  * 2mg of pure Simvastatin powder will be added to the 1:1:1 3Mix powder and will be stored together in an air tight porcelain container to avoid the exposure to moisture and light.
  * Upon clinical application the 3Mixtatin powder will be mixed with normal saline to form a paste and is then applied in the same manner as the Modified 3Mix-MP paste.
  Interventions: Drug: 3Mixtatin paste: Simvastatin mixed with modified triple antibiotic
- Group II Control group Modified triple antibiotic mix in propylene glycol (3Mix) (Active Comparator): * Removal of enteric coating/capsule of the three antibiotic tablets using a surgical blade.
  * 500 mg Metronidazole tab
  * 500 mg Ciprofloxacin tab
  * 200 mg Cefixime caps
  * Pulverization of each of the drug, will be done using a pestle & mortar, stored in an air tight porcelain container to avoid the exposure to moisture & light.
  * Pulverized powders will be stored at a temperature of 16°C.Powder should be allowed to be cooled to the room temperature before initiating the preparation of 3Mix-MP paste.
  * Powders will be mixed in the proportion of: 1:1:1 by volume (Hoshino et al., 1988).
  * Vehicle that will be used is Systane eye drops (Kharadly et al., 2022) it contains the two main components propylene Glycol (Macrogol) & polyethylene glycol.
  * The prepared antibiotic powder is mixed with the prepared vehicle in the ratio of 7:1 by volume. The two steps above are done after access cavity preparation to obtain a fresh mix.
  Interventions: Drug: 3Mix: Modified triple antibiotic mix in propylene glycol

INTERVENTIONS:
Drug: 3Mixtatin paste: Simvastatin mixed with modified triple antibiotic — * Drying the mucosa with gauze,topical anesthesia will be applied.
  * Administration of local anesthesia with vasoconstrictor.
  * Rubber dam isolation.
  * Caries removal & access cavity using a round bur mounted on a high-speed contra with coolant.
  * Removal of necrotic pulp tissue in coronal portion of the tooth using sharp excavator.
  * Radicular section will be kept untouched,no instrumentation.
  * Using disposable syringe Irrigation of the pulp chamber with 2.5% NaOCl.
  * In case of hemorrhage moist cotton immersed in 1% NaOCL will be placed to achieve hemostasis.
  * Drying the access cavity with sterile cotton pellets.
  * Freshly mixed 3Mix-MP or 3Mixtatin paste (according to group of intervention) will be transferred to the floor of the pulp chamber using an amalgam carrier & condensed over orifices using a moist cotton pellet.
  * Cavity sealing with RMGI capsules.
  * Same visit placement with preformed Stainless-steel crown(3M® ESPE)cemented with glass ionomer cement.
  Arms: (Group I Experimental Group):Simvastatin mixed with modified triple antibiotic (3Mixtatin)
Drug: 3Mix: Modified triple antibiotic mix in propylene glycol — * Drying the mucosa with gauze,topical anesthesia will be applied.
  * Administration of local anesthesia with vasoconstrictor.
  * Rubber dam isolation.
  * Caries removal & access cavity using a round bur mounted on a high-speed contra with coolant.
  * Removal of necrotic pulp tissue in coronal portion of the tooth using sharp excavator.
  * Radicular section will be kept untouched,no instrumentation.
  * Using disposable syringe Irrigation of the pulp chamber with 2.5% NaOCl.
  * In case of hemorrhage moist cotton immersed in 1% NaOCL will be placed to achieve hemostasis.
  * Drying the access cavity with sterile cotton pellets.
  * Freshly mixed 3Mix-MP or 3Mixtatin paste (according to group of intervention) will be transferred to the floor of the pulp chamber using an amalgam carrier & condensed over orifices using a moist cotton pellet.
  * Cavity sealing with RMGI capsules.
  * Same visit placement with preformed Stainless-steel crown(3M® ESPE)cemented with glass ionomer cement.
  Arms: Group II Control group Modified triple antibiotic mix in propylene glycol (3Mix)

SUMMARY:
This randomized clinical study aims to assess the clinical and radiographic success rate of the 3Mixtatin versus the 3Mix in LSTR in necrotic primary molars.

DETAILED DESCRIPTION:
Research question:

In necrotic primary molars with peri-radicular lesions and/or external root, resorption does adding Simvastatin to the triple antibiotic mix have higher clinical and radiographic success than the triple antibiotic paste solely?

Statement of the problem:

Primary teeth with necrotic pulp and extensive root resorption and/or furcal radiolucency are not uncommon scenarios that pediatric dentists are exposed to. Such clinical and radiographic presentations contraindicate the application of conventional pulpectomy treatment. Lesion Sterilization and Tissue Repair (LSTR) is an approach that has shown promising results in maintaining such teeth for up to 12 months. Primary teeth serve as a natural space maintainer, enable normal and healthy functioning of the child, and eliminate the chances for malocclusion and growth pattern disruptions. LSTR offers practitioners a promising option to save those teeth when all other treatment options seem impossible.

The Rationale for Conducting the Research:

In accordance to the popularity that LSTR has recently been gaining in the field of Pediatric dentistry, an abundance of studies have been conducted in the recent years. Researchers are striving to explore the plethora of possibilities and variances in the LSTR technique that could help clinicians practice better and achieve more for their patients. Amongst the alternatives is the recent and common detour towards regenerative dentistry.

Simvastatin, one of the materials, remains of high interest to the field due to its healing powers. However, to our knowledge insufficient studies are available on the direct comparison of the clinical and radiographic success including bone regeneration using the 3Mixtatin versus 3Mix alone. Furthermore, studies conducted warrant the need for further studies directly comparing 3Mixtatin with 3mix. Therefore, this study aims to come to a conclusion on whether the 3mix with the host's body defense and repair mechanism are sufficient to save a necrotic primary tooth or is some help in bone regeneration and healing promotion needed.

The LSTR technique involves non-instrumentation or minimal instrumentation followed by sterilization of the infected pulpal space by the placement of a triple antibiotic mixture in a propylene glycol vehicle to disinfect the microbial flora inhabiting the infected root canal systems and peri-apical lesions. The latter step achieves disinfection while tissue repair is then allowed to take place by the host's natural body defense mechanisms

The triple antibiotic paste (TAP/3mix), is an intracanal medicament that has continuously proven its efficacy and superiority for years against the microflora inhabiting necrotic canals predominantly Enterococcus Faecalis, the most prevalent organism in infected root canals. Metronidazole, ciprofloxacin, and minocycline, the oldest and most common combination suggested by Takushige et al., has been subjected to many studies and changes due to the discoloration caused by minocycline. As a result of, modified triple antibiotic paste (Modified-3mix) was introduced to replace minocycline with clindamycin.

Statins are antihyperlipidemic drugs, with a bio inductive feature that includes inhibition of bone resorption and promotion of osteoblast proliferation and differentiation as well as stimulating angiogenesis all of which aid in the healing process. In a clinical trial mixing modified 3mix with statins in, namely, Simvastatin; resulted in excellent clinical and radiographic success rates. Hence, modifying the LSTR technique to include regenerative materials such as statin is an extremely promising area of research.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 4-7 years.
* Positive parental informed consent.
* Restorable necrotic mandibular second primary molars with peri-radicular/furcal involvement and/or pathologic root resorption (external or internal).
* Presence of chronic apical abscess or sinus tract or furcation radiolucency. (Thakur et al., 2021)

Exclusion Criteria:

* Medically compromised children.
* Children with known allergy to any of the components being utilized.
* Molars near exfoliation.
* Molars with severely resorbed roots more than two thirds indicated for extraction
* Molars with insufficient coronal structure disabling proper coronal seal.
* Presence of periapical or interradicular radiolucent area which could compromise the permanent tooth bud. (Shetty et al., 2020)

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Absence of pathological mobility measured by (Miller's grades) | baseline
  Miller's Classification
  * Grade I: first distinguishable sign of movement
  * Grade II: movement of tooth which allows crown to deviate 1mm of its normal position
  * Grade III shows noticeable and increased movement of tooth more than 1mm in any direction or the tooth can be depressed into the socket.
  A reduction in grade of mobility from preoperative baseline will be considered as success while increased mobility will be recorded as failure
Absence of pathological mobility measured by (Miller's grades) | at 3 months post operative
  Miller's Classification
  * Grade I: first distinguishable sign of movement
  * Grade II: movement of tooth which allows crown to deviate 1mm of its normal position
  * Grade III shows noticeable and increased movement of tooth more than 1mm in any direction or the tooth can be depressed into the socket.
  A reduction in grade of mobility from preoperative baseline will be considered as success while increased mobility will be recorded as failure
Absence of pathological mobility measured by (Miller's grades) | at 6 months post operative
  Miller's Classification
  * Grade I: first distinguishable sign of movement
  * Grade II: movement of tooth which allows crown to deviate 1mm of its normal position
  * Grade III shows noticeable and increased movement of tooth more than 1mm in any direction or the tooth can be depressed into the socket.
  A reduction in grade of mobility from preoperative baseline will be considered as success while increased mobility will be recorded as failure
Absence of pathological mobility measured by (Miller's grades) | at 12 months post operative
  Miller's Classification
  * Grade I: first distinguishable sign of movement
  * Grade II: movement of tooth which allows crown to deviate 1mm of its normal position
  * Grade III shows noticeable and increased movement of tooth more than 1mm in any direction or the tooth can be depressed into the socket.
  A reduction in grade of mobility from preoperative baseline will be considered as success while increased mobility will be recorded as failure
Absence of post-operative pain (binary) | baseline
  Measured by asking the patient to identify presence or absence of pain
Absence of post-operative pain (binary) | at 3 months post operative
  Measured by asking the patient to identify presence or absence of pain
Absence of post-operative pain (binary) | at 6 months post operative
  Measured by asking the patient to identify presence or absence of pain
Absence of post-operative pain (binary) | at 12 months post operative
  Measured by asking the patient to identify presence or absence of pain
Absence of soft tissue pathologies (binary) | baseline
  Binary outcome measured visually by intraoral/extraoral examination
Absence of soft tissue pathologies (binary) | at 3 months post operative
  Binary outcome measured visually by intraoral/extraoral examination
Absence of soft tissue pathologies (binary) | at 6 months post operative
  Binary outcome measured visually by intraoral/extraoral examination
Absence of soft tissue pathologies (binary) | at 12 months post operative
  Binary outcome measured visually by intraoral/extraoral examination
Absence of pain on percussion (binary) | baseline
  Binary outcome measured by gentle tapping using the back of the mirror on the tooth
Absence of pain on percussion (binary) | at 3 months post operative
  Binary outcome measured by gentle tapping using the back of the mirror on the tooth
Absence of pain on percussion (binary) | at 6 months post operative
  Binary outcome measured by gentle tapping using the back of the mirror on the tooth
Absence of pain on percussion (binary) | at 12 months post operative
  Binary outcome measured by gentle tapping using the back of the mirror on the tooth

SECONDARY OUTCOMES:
Status of radiolucency if present at the periapical or at furcation area | baseline
  Comparison between pre-operative radiolucency and at follow up periods post-operatively to asses bone regeneration. Results will be recorded as Static-Increased-Decreased using customized stent for xray and Digora software for measurements.
Status of radiolucency if present at the periapical or at furcation area | at 6 months post operative
  Comparison between pre-operative radiolucency and at follow up periods post-operatively to asses bone regeneration. Results will be recorded as Static-Increased-Decreased using customized stent for xray and Digora software for measurements.
Status of radiolucency if present at the periapical or at furcation area | at 12 months post operative
  Comparison between pre-operative radiolucency and at follow up periods post-operatively to asses bone regeneration. Results will be recorded as Static-Increased-Decreased using customized stent for xray and Digora software for measurements.
Absence of external or internal root resorption | baseline , 6 ,12 months
  Binary outcome measured by comparing pre-operative x-ray with baseline and follow up x-rays. using customized stent

CONTACTS AND LOCATIONS:
Overall Officials: Rania Nasr, Professor, Study Director — Professor of pediatric dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chak RK, Singh RK, Mutyala J, Killi NK. Clinical Radiographic Evaluation of 3Mixtatin and MTA in Primary Teeth Pulpotomies: A Randomized Controlled. Int J Clin Pediatr Dent. 2022;15(Suppl 1):S80-S86. doi: 10.5005/jp-journals-10005-2216. PMID 35645497
- [Background] Hoshino E, Kurihara-Ando N, Sato I, Uematsu H, Sato M, Kota K, Iwaku M. In-vitro antibacterial susceptibility of bacteria taken from infected root dentine to a mixture of ciprofloxacin, metronidazole and minocycline. Int Endod J. 1996 Mar;29(2):125-30. doi: 10.1111/j.1365-2591.1996.tb01173.x. PMID 9206436
- [Background] Hoshino E, Kota K, Sato M, Iwaku M. Bactericidal efficacy of metronidazole against bacteria of human carious dentin in vitro. Caries Res. 1988;22(5):280-2. doi: 10.1159/000261121. PMID 3052845
- [Background] Aminabadi NA, Huang B, Samiei M, Agheli S, Jamali Z, Shirazi S. A Randomized Trial Using 3Mixtatin Compared to MTA in Primary Molars with Inflammatory Root Resorption: A Novel Endodontic Biomaterial. J Clin Pediatr Dent. 2016;40(2):95-102. doi: 10.17796/1053-4628-40.2.95. PMID 26950808
- [Background] Sain S, J R, S A, George S, S Issac J, A John S. Lesion Sterilization and Tissue Repair-Current Concepts and Practices. Int J Clin Pediatr Dent. 2018 Sep-Oct;11(5):446-450. doi: 10.5005/jp-journals-10005-1555. Epub 2018 Oct 1. PMID 30787561
- [Background] Takushige T, Cruz EV, Asgor Moral A, Hoshino E. Endodontic treatment of primary teeth using a combination of antibacterial drugs. Int Endod J. 2004 Feb;37(2):132-8. doi: 10.1111/j.0143-2885.2004.00771.x. PMID 14871180
- [Background] Thakur S, Deep A, Singhal P, Chauhan D. A randomized control trial comparing the efficacy of 3Mixtatin and Modified 3Mix-MP paste using lesion sterilization and tissue repair technique to conventional root canal treatment in primary molars of children aged 4-8 years: An in vivo study. Dent Res J (Isfahan). 2021 Nov 22;18:93. doi: 10.4103/1735-3327.330874. eCollection 2021. PMID 35003558